CLINICAL TRIAL: NCT06161207
Title: Prospective Randomized Controlled Trials on Clinical Outcomes of Indocyanine Green Tracer Using in 3D Plus Ultra High Resolution Laparoscopic Gastrectomy With Lymph Node Dissection for Locally Advanced Gastric Cancer
Brief Title: 3D-4K-ICG Laparoscopic Gastrectomy for Gastric Cancer
Acronym: 3D-4K-ICG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-31
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer; Surgery
Keywords: Indocyanine Green Tracer; Laparoscopic Gastrectomy; Gastric Cancer; Ultra High Resolution; 3D
MeSH Terms: conditions — Stomach Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3D-4K-ICG (Experimental): Indocyanine Green Tracer Using in 3D plus Ultra High Resolution Laparoscopic Gastrectomy with Lymph Node Dissection
  Interventions: Procedure: Indocyanine Green Tracer Using in 3D plus Ultra High Resolution Laparoscopic Gastrectomy with Lymph Node Dissection
- 4K-ICG (Experimental): Indocyanine Green Tracer Using in Ultra High Resolution Laparoscopic Gastrectomy with Lymph Node Dissection
  Interventions: Procedure: Indocyanine Green Tracer Using in 3D plus Ultra High Resolution Laparoscopic Gastrectomy with Lymph Node Dissection
- 3D (Placebo Comparator): 3D Laparoscopic Gastrectomy with Lymph Node Dissection
  Interventions: Procedure: Indocyanine Green Tracer Using in 3D plus Ultra High Resolution Laparoscopic Gastrectomy with Lymph Node Dissection

INTERVENTIONS:
Procedure: Indocyanine Green Tracer Using in 3D plus Ultra High Resolution Laparoscopic Gastrectomy with Lymph Node Dissection — Indocyanine green tracer is used with 3D plus ultra high resolution laparoscopic gastrectomy with lymph node Dissection for gastric cancer

SUMMARY:
Patients with locally advanced gastric adenocarcinoma (CT2-4a N-/+ M0) were selected as study subjects to investigate the safety, efficacy, and feasibility of ICG near-infrared imaging tracing in 3D plus ultra high resolution laparoscopic gastrectomy with lymph node dissection for gastric cancer.

DETAILED DESCRIPTION:
1. Research purpose: Patients with locally advanced gastric adenocarcinoma (CT2-4a N-/+ M0) were selected as study subjects to investigate the safety, efficacy, and feasibility of ICG near-infrared imaging tracing in 3D plus ultra high resolution laparoscopic gastrectomy with lymph node dissection for gastric cancer.
2. Research design: Prospective, single-center, randomized controlled, open-control, parallel assignment, superiority test.

2.1 Case group Group A (Study Group 1, 234 cases): ICG near-infrared imaging tracing in 3D plus ultra high resolution laparoscopic gastrectomy with lymph node dissection; Group B (Study Group 2, 234 cases): ICG near-infrared imaging tracing in ultra high resolution laparoscopic gastrectomy with lymph node dissection; Group C (Control Group 2, 234 cases) 3D laparoscopic gastrectomy with lymph node dissection

2.2 Estimate Sample Size The three-year disease-free survival (DFS) was the main effectiveness evaluation index in this study. The study implemented a superiority test (unilateral), assuming that both the study group's three-year DFS would be better than that of control group, according to previous research results of laparoscopic surgery for locally advanced GC in which the three-year DFS was 65.2%; therefore, the 3-year DFS of the control group would be 65.2%, assuming that the 3-year DFS of the experimental group could be increased by 12% to 77.2%. With an inspection level 0.0125 (unilateral) and an inspection efficiency of 0.8 and using PASS 11 log-rank tests (Lakatos) [Proportion surviving] the calculated sample size was N=211; namely, each group needed 211 people, considering cases of possible exclusion and loss to follow-up (10% drop out rate). The final sample size for each group was 234 cases, for a total of 702 cases.

2.3 randomization After laparoscopic exploration and confirmation that the cases complied with the standards, they were included in the randomized groups in this study. SAS 9.2 was used to produce a serial number ranging from 0001 - 702 corresponding to the treatment allocation, which was reserved in the data center and research center.

2.4 Blinding Method: This research adopts an open design.

2.5 Research cycle: Estimated enrollment cycle: complete enrollment within 2 years. Follow-up period: the enrollment of the first case was the starting point for follow-up. And the enrollment of last case to the postoperative pathology report (generally 2 weeks after surgery) was the endpoint of follow-up for secondary outcomes. Three years after the last case was enrolled was the follow-up endpoint for the main outcomes.

Estimated time: 2023.12-2025.12 (complete enrollment) to 2028.12 (complete follow-up)

Study Objects All patients who meet the inclusion criteria and do not conform to the exclusion criteria are qualified for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. cT2-4a, N-/+, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual, 8th Edition
4. No distant metastasis, no direct invasion of pancreas, spleen or other adjacent organs in the preoperative examinations
5. Performance status of 0 or 1 on the ECOG (Eastern Cooperative Oncology Group) scale
6. ASA (American Society of Anesthesiology) class I to III
7. Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous upper abdominal surgery (except for laparoscopic cholecystectomy)
4. History of previous gastric surgery (including ESD/EMR for gastric cancer)
5. Enlarged or bulky regional lymph node (diameter over 3cm) supported by preoperative imaging
6. Other malignant disease within the past 5 years
7. History of previous neoadjuvant chemotherapy or radiotherapy
8. History of unstable angina or myocardial infarction within past six months
9. History of cerebrovascular accident within past six months
10. History of continuous systematic administration of corticosteroids within one month
11. Requirement for simultaneous surgery for other disease
12. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
13. FEV1 (forced expiratory volume in one second)<50% of predicted values
14. Diffuse invasive gastric cancer
15. History of an iodine allergy
16. Patients who declined laparoscopic surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 3 years
  Disease-free survival is calculated from the day of surgery to the day of recurrence or death

SECONDARY OUTCOMES:
Operation time | 1 day
  Operation time
Total number of retrieved lymph nodes | 1 day
  Total number of retrieved lymph nodes
Noncompliance rate of lymph node dissection | 1 day
  Noncompliance rate of lymph node dissection
Relationship between fluorescent lymph nodes in group A and total number of lymph nodes in group A | 1 day
  Relationship between fluorescent lymph nodes in group A and total number of lymph nodes in group A
Relationship between fluorescent lymph nodes in Group A and positive lymph nodes in Group A (positive rate) | 1 day
  Relationship between fluorescent lymph nodes in Group A and positive lymph nodes in Group A (positive rate)
Relationship between fluorescent lymph nodes in Group A and negative lymph nodes in Group A (false positive rate) | 1 day
  Relationship between fluorescent lymph nodes in Group A and negative lymph nodes in Group A (false positive rate)
Relationship between non-fluorescent lymph nodes in Group A and negative lymph nodes in group A (negative rate) | 1 day
  Relationship between non-fluorescent lymph nodes in Group A and negative lymph nodes in group A (negative rate)
Relationship between nonfluorescent lymph nodes in Group A and positive lymph nodes in Group A (false negative rate) | 1 day
  Relationship between nonfluorescent lymph nodes in Group A and positive lymph nodes in Group A (false negative rate)
Relationship between fluorescent lymph nodes in group B and total number of lymph nodes in group B | 1 day
  Relationship between fluorescent lymph nodes in group B and total number of lymph nodes in group B
Relationship between fluorescent lymph nodes in Group B and positive lymph nodes in Group B (positive rate) | 1 day
  Relationship between fluorescent lymph nodes in Group B and positive lymph nodes in Group B (positive rate)
Relationship between fluorescent lymph nodes in Group B and negative lymph nodes in Group B (false positive rate) | 1 day
  Relationship between fluorescent lymph nodes in Group A and negative lymph nodes in Group A (false positive rate)
Relationship between non-fluorescent lymph nodes in Group B and negative lymph nodes in group B (negative rate) | 1 day
  Relationship between non-fluorescent lymph nodes in Group B and negative lymph nodes in group B (negative rate)
Relationship between nonfluorescent lymph nodes in Group B and positive lymph nodes in Group B (false negative rate) | 1 day
  Relationship between nonfluorescent lymph nodes in Group B and positive lymph nodes in Group B (false negative rate)
Number of metastatic lymph nodes | 1 day
  Number of metastatic lymph nodes
Metastasis rate of lymph nodes | 1 day
  Metastasis rate of lymph nodes
Morbidity and mortality rates | 30 day
  Morbidity and mortality rates
3-year overall survival rate | 3 years
  3-year overall survival rate
3-year recurrence pattern | 3 years
  3-year recurrence pattern
Postoperative recovery course | 30 days
  Postoperative recovery course
Intraoperative situation | 30 days
  Intraoperative situation
Postoperative nutritional status | 3 years
  Postoperative nutritional status
Inflammatory and immune response | 30 days
  Inflammatory and immune response
Postoperative quality of life (measured by EQ-5D) | preoperative, postoperative 1 month and postoperative 1 year
  Postoperative quality of life (measured by EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-ming Huang, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No